CLINICAL TRIAL: NCT02944487
Title: A Randomised, Double-blind, Placebo-controlled Ascending Dose Tolerance Study of OGT 923 in Healthy Male Volunteers
Brief Title: A Study to Assess the Safety and Pharmacokinetics of Lucerastat (OGT 923) in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: OGT923-001
Record Dates: First submitted 2016-10-24; First posted 2016-10-26 (Estimated); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Healthy Subjects
Keywords: safety; pharmacokinetics
MeSH Terms: interventions — migalastat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Single ascending doses of lucerastat (Experimental): Subjects were enrolled sequentially in 4 groups and received a single oral dose of lucerastat from 100 mg to 1000 mg in the morning of Day 1
  Interventions: Drug: Lucerastat
- B.i.d. Dose Group (Experimental): Subjects received two doses of lucerastat (2 x 1 g) 12 hours apart on Day 1
  Interventions: Drug: Lucerastat
- Placebo for singe ascending doses (Placebo Comparator): These subjects received matching placebo administered orally in the morning of Day 1
  Interventions: Drug: Placebo
- Placebo for b.i.d.Group (Placebo Comparator): These subjects received matching placebo administered orally in the morning and in the evening of Day 1
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lucerastat — Hard gelatin capsule for oral administration containing lucerastat
  Other Names: OGT-923; ACT-434964
  Arms: B.i.d. Dose Group; Single ascending doses of lucerastat
Drug: Placebo — Matching placebo capsules
  Arms: Placebo for b.i.d.Group; Placebo for singe ascending doses

SUMMARY:
The objectives of this study were to evaluate the safety and tolerability of lucerastat, and to determine its pharmacokinetic profile as single oral doses at different strengths.

DETAILED DESCRIPTION:
The subjects were enrolled sequentially to five dose groups, starting with the lowest dose level. Subjects could participate in only one Group.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form.
* Male subjects aged from 18 to 45 years at screening.
* Body weight between 50 and 100 kg and body mass index (BMI) between 18.0 and 29.0 kg/m2 at screening.
* Healthy on the basis of physical examination, cardiovascular assessments and laboratory tests.

Exclusion Criteria:

* History or clinical evidence of any disease or medical / surgical condition or treatment, which may put the subject at risk of participation in the study or may interfere with the absorption, distribution, metabolism or excretion of the study treatments.
* Serious adverse reaction or hypersensitivity to any drug.
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2002-10; Primary Completion 2002-12 (Actual); Study Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events (AEs) | From baseline up to 7 days post-administration
  An AE was defined as any untoward medical occurrence in a clinical investigation subject, which did not necessarily have a causal relationship with the treatment.
Maximum plasma concentration (Cmax) of lucerastat after single ascending doses of lucerastat | PK Blood samples were collected at pre-dose and at scheduled time points up to 24 hours post administration
  Cmax was determined directly from the observed plasma concentration-time curves of lucerastat in subjects receiving a single dose.
Maximum plasma concentration (Cmax) of lucerastat after two daily doses of lucerastat | PK Blood samples were collected at pre-dose and at scheduled time points up to 48 hours after the first administration
  Cmax was determined directly from the observed plasma concentration-time curves of lucerastat in subjects receiving lucerastat twice daily.
Time to reach Cmax (tmax) of lucerastat after single ascending doses of lucerastat | PK Blood samples were collected at pre-dose and at scheduled time points up to 24 hours post administration
  tmax was determined directly from the observed plasma concentration-time curves of lucerastat in subjects receiving a single dose.
Time to reach Cmax (tmax) of lucerastat after two daily doses of lucerastat | PK Blood samples were collected at pre-dose and at scheduled time points up to 48 hours after the first administration
  tmax was determined directly from the observed plasma concentration-time curves of lucerastat in subjects receiving lucerastat twice daily.
Area under the plasma concentration-time curves (AUC) of lucerastat after single ascending doses of lucerastat | PK Blood samples were collected at pre-dose and at scheduled time points up to 24 hours post administration
  AUC was calculated from time zero to time t (last PK blood sample in which drug was detected) and extrapolated to infinity for subjects receiving a single dose.
Area under the plasma concentration-time curves (AUC) of lucerastat after two daily doses of lucerastat | PK Blood samples were collected at pre-dose and at scheduled time points up to 48 hours after the first administration
  AUC was calculated from time zero to time t (last PK blood sample in which drug was detected) and extrapolated to infinity for subjects receiving lucerastat twice daily
Terminal elimination half-life (t1/2) of lucerastat after single ascending doses of lucerastat | PK Blood samples were collected at pre-dose and at scheduled time points up to 24 hours post administration
  t1/2 was calculated from the corresponding plasma concentrations-time curves for subjects receiving a single dose
Terminal elimination half-life (t1/2) of lucerastat after two daily doses of lucerastat | PK Blood samples were collected at pre-dose and at scheduled time points up to 48 hours after the first administration
  t1/2 was calculated from the plasma concentrations-time curves for subjects receiving lucerastat twice daily

SECONDARY OUTCOMES:
Change from baseline in heart rate | Up to 24 hours post administration
Change from baseline in blood pressure | Up to 24 hours post administration
Change from baseline in electrocardiogram (ECG) variables | Up to 24 hours post administration
Change from baseline in laboratory tests | Up to 24 hours post administration

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Idorsia Pharmaceuticals
Locations (1):
- Investigator Site, Tranent, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guerard N, Morand O, Dingemanse J. Lucerastat, an iminosugar with potential as substrate reduction therapy for glycolipid storage disorders: safety, tolerability, and pharmacokinetics in healthy subjects. Orphanet J Rare Dis. 2017 Jan 14;12(1):9. doi: 10.1186/s13023-017-0565-9. PMID 28088251